CLINICAL TRIAL: NCT06008275
Title: Pilot Clinical Trial Examining the Safety and Efficacy of Neratinib in Combination With Ruxolitinib in Patients With Chemotherapy-pretreated Metastatic Triple Negative Breast Cancer With Chest Wall Recurrence
Brief Title: Neratinib in Combination With Ruxolitinib in Patients With mTNBC
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 023-340
Record Dates: First submitted 2023-08-18; First posted 2023-08-23 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Triple-Negative Breast Carcinoma; Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — neratinib; ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- neratinib + ruxolitinib (Experimental): There is only one arm
  Interventions: Drug: Neratinib Oral Tablet; Drug: Ruxolitinib Oral Tablet

INTERVENTIONS:
Drug: Neratinib Oral Tablet — 240mg oral daily. Dosing will follow standard dose escalation procedures
Drug: Ruxolitinib Oral Tablet — 20mg oral twice daily. Dosing will follow standard initial dose recommendation procedure
  Other Names: Jakafi

SUMMARY:
The goal of this clinical trial is to assess the safety and efficacy of combined ruxolitinib and neratinib in patients with chemotherapy-pretreated metastatic triple negative breast cancer. This trial will evaluate one dosing schedule of neratinib in ruxolitinib in patients with metTNBC with locoregional recurrence.

DETAILED DESCRIPTION:
Metastatic triple negative breast cancer (metTNBC) lacks expression of estrogen receptor (ER), progesterone receptor (PR), and human epidermal growth factor receptor 2 (HER2), making it unresponsive to both endocrine and HER2-targeted therapies. Chest wall recurrence is common in patients with treatment resistant metTNBC and leads to substantial morbidity as no successful therapeutic options exist. Patients suffer with escalated progression of disease across the entire chest wall with substantial wound control issues. Chest wall recurrence generally occurs within one year following chemotherapy or immunotherapy given with curative intent, and in general signifies metTNBC that is primary resistant to standard therapy.

There is long standing evidence that EGFR is an important signaling pathway in metTNBC as this cancer overexpresses EGFR compared to other breast cancer subtypes. This exposes a pathway that is targetable for treatment, making EGFR a compelling molecular therapeutic target in metTNBC. Another key contributor to progression of TNBC is the JAK/STAT3 signaling pathway and assessments of EGFR have shown that it is a positive regulator of STAT3 that drives proliferation and survival of metTNBC.

The investigators hypothesize that combined inhibition of EGFR and JAK/STAT3 using neratinib and ruxolitinib will lead to greater inhibition of the critically important EGFR pathway in TNBC with greater efficacy than targeting EGFR or JAK/STAT3 alone.

ELIGIBILITY:
Inclusion Criteria:

* A patient will be considered for enrollment in this study if all the following criteria are met:

  1. Female patients ≥18 years of age
  2. Have a diagnosis of metastatic TNBC previously treated with standard anthracycline, cyclophosphamide, and taxane chemotherapy, unless there was a contraindication to doxorubicin, in which case prior treatment with this agent is not required.

     Note. TNBC defined as ER-negative tumors with ≤10% tumor nuclei immunoreactivity, or "ER Low Positive" as defined by the updated ASCO/CAP guidelines 2020.
  3. Have not received more than 4 prior chemotherapy regimens for metastatic disease. Prior platinum and/or taxane therapy in the adjuvant or metastatic setting is permitted. Patients with more than 4 prior regimens may be allowed on study per physician discretion, if ECOG PS is 0-1.
  4. Have locoregional (e.g., breast, chest wall, regional lymphatic) or pulmonary or hepatic metastatic disease that is amenable to core needle biopsy. If a research biopsy from a patient's metastatic disease cannot be safely obtained, a skin biopsy is permitted. If a skin biopsy cannot be safely obtained, patients may still be eligible, per physician discretion.
  5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
  6. Have adequate hematologic function, defined by:

     1. Absolute neutrophil count (ANC) >1500/µL
     2. Platelet count ≥100,000/ µL
     3. Hemoglobin ≥9 g/dL or ≥5.6 mmol/L
  7. Have adequate liver function, defined by:

     1. AST and ALT ≤2.5 x the upper limit of normal (ULN) or ≤5 x ULN in presence of liver metastases
     2. Total bilirubin ≤1.5 x ULN OR direct bilirubin ≤ULN for patients with total bilirubin levels >1.5 × ULN
  8. Have adequate renal function, defined by:

     a. Serum creatinine ≤1.5 x ULN or calculated creatinine clearance of ≥30 mL/min
  9. Patients who have a history of brain metastasis are eligible for the study provided that all the following criteria are met:
  10. Brain metastases which have been treated
  11. Off-treatment with steroids before administration of the first dose of treatment
  12. No ongoing requirement for dexamethasone or anti-epileptic drugs
  13. No clinical or radiological evidence of progression of brain metastases
  14. Patients must be accessible for treatment and follow-up.
  15. All patients must be able to understand the investigational nature of the study and give written informed consent prior to study entry.

Exclusion Criteria:

* A patient will be ineligible for inclusion in this study any of the following criteria are met:

  1. Has received a live vaccine or live-attenuated vaccine within 30 days of the first dose of study treatment. Administration of killed vaccines is allowed.
  2. Has peripheral neuropathy ≥grade 2
  3. Has completed previous radiotherapy for metastatic disease <2 weeks prior to study treatment initiation
  4. Has an active infection requiring systemic therapy
  5. Has significant cardiovascular disease, such as:

     1. History of myocardial infarction, acute coronary syndrome, or coronary angioplasty/stenting/bypass grafting within the last 6 months
     2. Congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV, or history of CHF NYHA class III or IV.
  6. Has a known history of active tuberculosis
  7. Women who are pregnant or lactating. All patients with reproductive potential must agree to use effective contraception from time of study entry until at least 3 months after the last administration of study drug.
  8. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation such as:

     1. severe impaired lung functions as defined as spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air
     2. liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).
  9. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's full participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the Treating Physician.
  10. Has received prior systemic anti-cancer therapy within 2 weeks prior to study treatment.
  11. Has received investigational agents within 4 weeks prior to study treatment. Monoclonal antibody agents should have a 4-week (28 day) washout period.
  12. Any other investigational or anti-cancer treatments while participating in this study
  13. Any other active malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 18 months
  Calculate objective response rate (CR+PR) associated with neratinib in combination ruxolitinib. Objective response rate will be calculated by defining the proportion of patients who have a complete or partial response to the study therapy, as determined by the treating physician.

SECONDARY OUTCOMES:
Duration of Response | 18 months
  Calculate duration of response associated with neratinib in combination with ruxolitinib. Duration of response will be calculated from the time of tumor response to disease progression in patients responding to study therapy

OTHER OUTCOMES:
Genetic Evaluation | 18 months
  Signaling signatures of research biopsies will be analyzed via Next Generation Sequencing and Reverse Phase Protein Array

CONTACTS AND LOCATIONS:
Overall Officials: Joyce A O'Shaughnessy, MD, Principal Investigator — Baylor Scott and White Research Institute
Locations (1):
- Baylor University Medical Center, Baylor Charles A Sammons Cancer Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided